CLINICAL TRIAL: NCT06315985
Title: The Effect of Classical Turkish Music on Stress and Sleep Quality in Pregnant Women Diagnosed With Preeclampsia in the Clinic
Brief Title: Classical Turkish Music for Pregnant Women With Preeclampsia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tarsus University (Other)
Responsible Party: Principal Investigator, Gulay Aksoy, Midwife, Student on master degree program at Tarsus University Midwifery Department, Tarsus University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GAksoy
Record Dates: First submitted 2024-03-12; First posted 2024-03-18 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Pre-Eclampsia
Keywords: Pre-Eclampsia; Classical Turkish Music; Sleep Quality; Stress
MeSH Terms: conditions — Pre-Eclampsia; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: This was a parallel group, randomized controlled trial conducted in a tertiary hospital in Mersin city center, Turkey. In parallel with the purpose of the study, participants were selected from the pregnant women diagnosed with preeclampsia who were hospitalized at Mersin City Training and Research Hospital.The population of the research is the G* Power 3.1.9.4 was determined by analysis using. In the analysis, the sample size was taken as a sample size of at least 80%, a medium effect size (0.5) and a two-way type 1 error value of 0.05, since no study similar to the study could be found, and a total of 128 pregnant women were included in the two groups (in each group) to determine the difference between the averages of two independent groups. It was calculated as 64 pregnant women). Considering the drop out rate of 10% during the research, the total number of samples was found to be 142 (experimental group: n=71, control group: n=71) pregnant women.
Who Masked: Participant
Masking Description: Participant will be masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): This was a parallel group, randomized controlled trial. Experimental Group will listen to the music for three days.
  Interventions: Other: Experimental group: Listenning to the Turkish Classical Music to pregnant women diagnosed with preeclampsia
- Control Group (No Intervention): Control Group will take routine care

INTERVENTIONS:
Other: Experimental group: Listenning to the Turkish Classical Music to pregnant women diagnosed with preeclampsia — The music to be used in the research will be applied together with midwifery practices and is not a treatment option, tool or treatment option for any disease. Although listening to Classical Turkish music has no effect on treatment and care, it does not have a harmful effect on pregnant women. The participant can withdraw from the study at any time without giving any reason. The Personal Information Form, Perceived Stress Scale, and Pittsburgh Sleep Quality Index (PSQI) will be administered to the pregnant women in both groups participating in the study by face-to-face interviews with the individuals on the first day of their admission to the clinic. At the end of the third day, the Perceived Stress Scale and Pittsburgh Sleep Quality Index (PSQI) scales will be re-administered to both groups.
  Other Names: Experimental group:
  Arms: Experimental Group

SUMMARY:
Stress and Sleep of Classical Turkish Music in Pregnant Women Diagnosed with Preeclampsia in Clinics The study to be carried out to determine the effect on quality is a randomized controlled experimental research. All patients who comply with the limitations of the study and volunteer will be included in the study. When the studies in the literature are examined, there are a limited number of studies on the effects of music on pregnant women diagnosed with preeclampsia, and no studies have been found on the effects of music on stress and sleep quality in pregnant women with preeclampsia. This research aimed to determine the effect of Classical Turkish Music on stress and sleep quality in pregnant women diagnosed with Preeclampsia in clinics.

DETAILED DESCRIPTION:
Pregnancy is a natural process that has physiological, psychological and sociological effects on women's lives and is special and important for every woman, affecting both the person and her family (Koyucu et al., 2020; Toker, 2018; Coşkun, 2016). Maternal age, number of pregnancies and births, adverse environmental conditions such as alcohol and cigarette use, radiation, malnutrition, diseases the woman has during the pre-pregnancy period or diseases that occur during pregnancy all negatively affect the health of the mother and the fetus, leading to a risky pregnancy. (Taşkın, 2016; Toker, 2018). According to Turkey Demographic and Health Survey 2018 (TNSA, 2018) data, when births occurring in Turkey are examined, it is seen that 65.7% are in any high risk category and 35% are in at least one inevitable high risk category (TNSA , 2018).

According to the report titled "Trends in Maternal Mortality" prepared by the World Health Organization (WHO), UNICEF, UNFPA, World Bank Group and UNDESA/Population Division; In 2020, an estimated 287,000 women per year worldwide died from preventable causes related to pregnancy and childbirth, approximately 800 every day; This means that one woman dies every two minutes (UNFPA, 2023; WHO, 2023; UNICEF, 2023; WHO, 2023). According to the 2020 data of the Ministry of Health, maternal mortality rates in our country decreased to 13.1 per hundred thousand as of 2019 (Ministry of Health, 2020).

10-15% of direct maternal deaths worldwide are related to preeclampsia and eclampsia, ranking 3rd among major complications (Akolekar et al., 2013; Demirci, 2022; WHO, 2020).

According to 2019 data in our country, the first four most common causes of maternal deaths are; cardiovascular diseases (29%), embolism (16.1%), hypertension (14.2%) and bleeding (10.3%) (Maternal deaths study report, 2021; Republic of Turkey Ministry of Health Health Statistics Yearbook, 2021) . According to 2022 data of the Turkish Gynecology and Obstetrics Association, it is estimated that at least 42,000 maternal deaths annually are caused by preeclampsia (Turkish Gynecology and Obstetrics Association, 2022).

Preeclampsia; It is a pregnancy-specific disease and is a symptom characterized by hypertension (systolic blood pressure 140 mmHg and above and/or diastolic blood pressure 90 mmHg and above) and end organ dysfunction with or without proteinuria after the 20th week of pregnancy (Jung and al., 2022). Preeclampsia is a disease whose physiopathology is still not fully known. The decline in prognosis with the disappearance of the placenta after birth indicates that preeclampsia may be of placental origin (Thilaganathan & Kalafat., 2019). Preeclampsia causes dysfunction in the liver, kidney, uterus, respiratory, cerebrovascular and cardiovascular systems. If it is not diagnosed at an early stage and appropriate treatment is not provided, it may become severe in a short time and turn into eclampsia. Eclampsia is a condition that occurs with the addition of convulsions in a pregnant woman with preeclampsia symptoms, without any neurological or metabolic disease (Hansson et al., 2015; Dag et al., 2015; Günkur, 2019; Akalın & Şahin, 2018).

Since preeclampsia is in the risk category during pregnancy, it may cause increased anxiety in pregnant women regarding birth and motherhood, as well as conditions such as stress and sleep disorders. In this context, the physiological health of the pregnant woman also negatively affects her psychosocial state. Hospitalization experience and bed rest in pregnant women with a risky pregnancy diagnosis such as preeclampsia; Reasons such as being away from family and home, activity limitation, uncertainty, being in an unknown environment, not being able to fulfill their roles, anxiety about the fetus and their own health, repeated laboratory and screening tests can cause stressful results (Gourounti et al., 2015; Özçetin & Erkan). , 2019).

In the studies carried out; It has been determined that the risk of IUGR increases in women with high stress levels during pregnancy, there is an increase in cortisol and adrenaline levels, there is a decrease in dopamine and serotonin levels, the fetus is more active, and mood and irregular sleep changes are experienced more frequently in the pregnant woman (Yousefzadeh, 2022; Spehar et al. ., 2018; Şen, 2020; Karadeniz et al., 2023). Again in the literature; It has been stated that in pregnant women hospitalized in clinics, insomnia complaints are common during hospitalization due to the treatment regimen and hospital conditions, and there is dissatisfaction with sleep quality (Spehar et al., 2018; Şen, 2020; Karadeniz et al., 2023). However, approximately 1/3 of human life is spent sleeping. Restricting sleep or reducing its quality are factors that can cause detrimental effects on life expectancy and quality (Ulusoy, 2020; Reutrakul & Van, 2018). With sleep problems during pregnancy; adverse perinatal outcomes such as increases in blood pressure,

Type of Research:

It was planned as a randomized controlled experimental study to determine the effect of Classical Turkish Music on Stress and Sleep Quality in Pregnant Women Diagnosed with Preeclampsia. All patients who comply with the limitations of the study and volunteer will be included in the study. The research is a cross-sectional study, and quantitative data will be collected using the online survey technique, one of the data collection methods.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women are hospitalized for three to five days with the diagnosis of Preeclampsia,
* No hearing problems (as music will be played),
* Having the appropriate level of consciousness,
* Must be at least literate (in order to obtain consent),
* Being over 18 years old (in order to obtain consent),
* No communication problems,
* Having a live fetus.
* Pregnant women who agree to participate in the research verbally and in writing will be included in the research.

Exclusion Criteria:

* Not agreeing to participate in the research verbally or in writing,
* Illiteracy,
* Not being under 18 years of age,
* Having a communication problem,
* Having a hearing problem,
* Being hospitalized for less than three days with a diagnosis of preeclampsia,
* Taking MgSO4
* Having previously been diagnosed with a sleep disorder
* Having a diagnosis of DM other than preeclampsia
* Being hospitalized for less than three days with a diagnosis of preeclampsia,
* The newborn is not healthy.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 142 (Estimated)
Dates: Start 2024-03-20 (Estimated); Primary Completion 2024-09-20 (Estimated); Study Completion 2025-03-20 (Estimated)

PRIMARY OUTCOMES:
Perceived Stress | 15-30 minutes
  It was developed by Cohen et al. in 1983, and Turkish validity and reliability studies were conducted by Erci in 2006. Perceived Stress Scale: 7 items containing positive statements (items 4-5-6-7-9-10 and 13) are scored in reverse and consists of 14 items in total. These items are scored by the individual on a 5-point Likert type scale (1=Never, 2=Almost never, 3=Sometimes, 4=Often, 5=Very often). The analysis of the scale is carried out on the total score. A high total score means a high Perceived Stress Level Scale. It can be said that participants whose score range is between 0-35 are at a positive stress level, can cope with stress effectively, and the coping mechanisms they use are functional. It can be said that the methods used by the participants with a score range between 36-56 are not functional and therefore they cannot cope with stress effectively.

SECONDARY OUTCOMES:
Sleep Quality | 15-30 minutes
  It was developed by Buyssee et al. in 1989 to evaluate sleep quality in clinical research and psychiatric practices, and its Turkish validity and reliability was confirmed by Ağargün et al. in 1996. PSQI is a 24-question index consisting of 20 questions valued from 0 to 3 and 4 open-ended questions. The patient answers 19 questions himself, while the patient's roommate or bedmate answers 5 questions. The 19 questions answered by the patient are evaluated in 7 categories and combined to obtain the PSQI global score, which ranges between 0 and 21. A total score from the scale greater than 5 is evidence of poor sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Gülay Aksoy, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gestational Hypertension and Preeclampsia: ACOG Practice Bulletin, Number 222. Obstet Gynecol. 2020 Jun;135(6):e237-e260. doi: 10.1097/AOG.0000000000003891. PMID 32443079
- [Background] Hypertension in pregnancy. Report of the American College of Obstetricians and Gynecologists' Task Force on Hypertension in Pregnancy. Obstet Gynecol. 2013 Nov;122(5):1122-1131. doi: 10.1097/01.AOG.0000437382.03963.88. No abstract available. PMID 24150027
- [Background] Chang SC, Chen CH. Effects of music therapy on women's physiologic measures, anxiety, and satisfaction during cesarean delivery. Res Nurs Health. 2005 Dec;28(6):453-61. doi: 10.1002/nur.20102. PMID 16287051
- [Background] Dag ZO, Isik Y, Turkel Y, Alpua M, Simsek Y. Atypical eclampsia and postpartum status epilepticus. Pan Afr Med J. 2015 Jan 7;20:17. doi: 10.11604/pamj.2015.20.17.5831. eCollection 2015. PMID 25995814
- [Background] Hansson SR, Naav A, Erlandsson L. Oxidative stress in preeclampsia and the role of free fetal hemoglobin. Front Physiol. 2015 Jan 13;5:516. doi: 10.3389/fphys.2014.00516. eCollection 2014. PMID 25628568
- [Background] Jung E, Romero R, Yeo L, Gomez-Lopez N, Chaemsaithong P, Jaovisidha A, Gotsch F, Erez O. The etiology of preeclampsia. Am J Obstet Gynecol. 2022 Feb;226(2S):S844-S866. doi: 10.1016/j.ajog.2021.11.1356. PMID 35177222
- [Background] Reutrakul S, Van Cauter E. Sleep influences on obesity, insulin resistance, and risk of type 2 diabetes. Metabolism. 2018 Jul;84:56-66. doi: 10.1016/j.metabol.2018.02.010. Epub 2018 Mar 3. PMID 29510179
- [Background] Spehar SM, Mission JF, Amanda Shupe, Facco FL. Prolonged antepartum hospitalization: no time for rest. J Perinatol. 2018 Sep;38(9):1151-1156. doi: 10.1038/s41372-018-0155-2. Epub 2018 Jul 9. PMID 29983417
- [Background] Thilaganathan B, Kalafat E. Cardiovascular System in Preeclampsia and Beyond. Hypertension. 2019 Mar;73(3):522-531. doi: 10.1161/HYPERTENSIONAHA.118.11191. PMID 30712425
- [Background] Yang M, Li L, Zhu H, Alexander IM, Liu S, Zhou W, Ren X. Music therapy to relieve anxiety in pregnant women on bedrest: a randomized, controlled trial. MCN Am J Matern Child Nurs. 2009 Sep-Oct;34(5):316-23. doi: 10.1097/01.NMC.0000360425.52228.95. PMID 19713801
- [Background] Akolekar R, Syngelaki A, Poon L, Wright D, Nicolaides KH. Competing risks model in early screening for preeclampsia by biophysical and biochemical markers. Fetal Diagn Ther. 2013;33(1):8-15. doi: 10.1159/000341264. Epub 2012 Aug 16. PMID 22906914
- See also: Gourounti C, Karpathiotaki N, Vaslamatzis G. Psychosocial stress in high risk pregnancy. Int Arch Med. 2015;8:1-9. — https://dergipark.org.tr/en/download/article-file/809241
- See also: United Nations Population Fund, 2023, Trends in Maternal Mortality 2000-2020, Estşmates by WHO, UNİCEF, UNFPA, World Bank Group and UNDESA/ Population Division — https://www.unfpa.org/publications/trends-maternal-mortality-2000-2020
- See also: WHO, 2020 — https://www.who.int/news-room/fact-sheets/detail/maternal-mortality
- See also: World Health Organization, 2023, Trends in maternal mortality 2000 to 2020: estimates by WHO, UNICEF, UNFPA, World Bank Group and UNDESA/Population Division — https://www.who.int/publications/i/item/9789240068759
- See also: World Health Organization, UNICEF, United Nations Population Fund and The World Bank, Trends in Maternal Mortality: 2000 to 2020 WHO, Geneva, 2023. — https://www.who.int/publications/i/item/9789240068759
- See also: Yüksekol, Ö. D., & Başer, M. (2020). Preeklampsili Gebelerde Tamamlayıcı Ve Bütünleşik Terapilerin Kullanımı. Turkish Journal of Science and Health, 1(2), 79-83 — https://dergipark.org.tr/en/download/article-file/1178083
- See also: Yousefzadeh, 2022; Covıd-19 Pandemisinin Gebelikte Stres Ve Yaşam Kalitesi Üzerine Etkisi, Yükseklisans Tezi — https://tez.yok.gov.tr/UlusalTezMerkezi/tezSorguSonucYeni.jsp
- See also: Yeten, H. U. (2023). Müziğin geçiş fazı ve sonrası doğum sürecine etkisinin incelenmesi (Master's thesis, Biruni Üniversitesi). — https://openaccess.biruni.edu.tr/xmlui/handle/20.500.12445/3497
- See also: Yalçın, A., & Saygın, M. (2021). Koku ve Uyku Kalitesi İlişkisinin Araştırılması. Uyku Bülteni, 2(2), 38-48.) — https://dergipark.org.tr/en/download/article-file/1544747
- See also: Ulusoy, Y. (2020). Uykunun Egzersiz Performansı Üzerine Etkisi-Uyku, Beslenme ve Toparlanma İlişkisi. Çanakkale Onsekiz Mart Üniversitesi Spor Bilimleri Dergisi, 3(3), 1-22. — https://dergipark.org.tr/en/download/article-file/1381618
- See also: Türkiye Ulusal Anne Ölümleri Çalışması, 2005 — https://fs.hacettepe.edu.tr/hips/dosyalar/Ara%C5%9Ft%C4%B1rmalar%20-%20raporlar/Di%C4%9Fer%20Ara%C5%9Ft%C4%B1rmalar/UAOC2005-AnaRapor.pdf
- See also: Türkiye Anne Ölümleri Raporu 2015-2019 — https://hsgm.saglik.gov.tr/depo/Yayinlarimiz/Raporlar/Turkiye_Anne_Olumleri_Raporu_2015-2019.pdf
- See also: TNSA, 2018 — http://www.sck.gov.tr/wp-content/uploads/2020/08/TNSA2018_ana_Rapor.pdf
- See also: T.C. Sağlık Bakanlığı Sağlık İstatistikleri Yıllığı 2021 — https://dosyasb.saglik.gov.tr/Eklenti/45316/0/siy2021-turkcepdf.pdf
- See also: .C. Sağlık Bakanlığı Halk Sağlığı Genel Müdürlüğü Kadın ve Üreme Sağlığı Dairesi Başkanlığı Ankara-2021 Anne Ölümleri Raporu — https://sbsgm.saglik.gov.tr/Eklenti/45316/0/siy2021-turkcepdf.pdf
- See also: Şen, G. (2020). Gebelikte Görülen Yakınmaların Uyku Kalitesine Etkisi. — https://tez.yok.gov.tr/UlusalTezMerkezi/tezSorguSonucYeni.jsp
- See also: Şası, G. (2020), Doğum Korkusu ve Ağrısının Azaltılmasında Müziğin Etkisi, Yüksek Lisans Tezi, Marmara Üniversitesi Sağlık Bilimleri Enstitüsü, Ebelik Anabilim Dalı, İstanbul, — https://tez.yok.gov.tr/UlusalTezMerkezi/tezDetay.jsp?id=bmsys4bz_WeKQijisRncCw&no=kA8QX8tlS-sPSO58z-EIZg
- See also: Santur, S. G., & Özşahin, Z. (2021). Kadın hayatının evrelerinde uyku ve ebelik yaklaşımı. The Journal of Turkish Family Physician, 12(4), 207-216. — http://turkishfamilyphysician.com/makaleler/derleme/kadin-hayatinin-evrelerinde-uyku-ebelik-yaklasimi/
- See also: Özçetin, Y. S. Ü., & Erkan, M. (2019). Yüksek riskli gebelerde psikolojik sağlamlık, algılanan stres ve psikososyal sağlık. Cukurova Medical Journal, 44(3), 1017-1026. — https://dergipark.org.tr/tr/download/article-file/809241
- See also: Koyucu, R. G., Ülkar, D., & Erdem, B. (2020). Primipar Ve Multipar Gebelerin Gebelik Streslerinin Karşılaştırılması. İnönü Üniversitesi Sağlık Hizmetleri Meslek Yüksek Okulu Dergisi, 8(3), 652-663.) — https://dergipark.org.tr/tr/download/article-file/1126933
- See also: Karamızrak, N. (2019). Kardiyovasküler Hastalıklarda Müzik ile Terapi. Koşuyolu Heart Journal, 22(2), 120- 125 — https://dergipark.org.tr/tr/download/article-file/785904
- See also: Karadeniz, M., Ser, M. H., & Şenel, G. B. (2023). Gebelikte Uyku Kalitesinin Trimesterlere Göre Değerlendirilmesi ve İlişkili Faktörlerin İncelenmesi. Journal of Turkish Sleep Medicine, 10(2). — https://cms.jtsm.org/Uploads/Article_60444/JTSM-10-116.pdf
- See also: Günkur, K. (2019). Preeklampside Trombosit Aktive Edici Faktör Asetil Hidrolaz, Paraoksonaz, Myeloperoksidaz ile Serum Amiloid A Düzeylerinin Belirlenmesi ve Aralarındaki İlişkinin İncelenmesi (Master's thesis, Sağlık Bilimleri Enstitüsü). — https://acikbilim.yok.gov.tr/bitstream/handle/20.500.12812/101849/yokAcikBilim_10085075.pdf?sequence=-1&isAllowed=y
- See also: Gülay, K. U. R. T., Hüsniye, D. İ. N. Ç., & Günaydın, S. Gebelikte Ve Doğum Ağrısının Kontrolünde Müzikoterapinin Kullanımı. Kırşehir Ahi Evran Üniversitesi Sağlık Bilimleri Dergisi, 1(3), 194-199. — https://dergipark.org.tr/en/download/article-file/1884484
- See also: Demirci, G. (2022). Preeklampside anne ve kord kanında netrin-1 düzeylerinin incelenmesi ve bunların vitamin D, vitamin B12, folik asit ile ilişkisinin araştırılması. — https://gcris.pau.edu.tr/bitstream/11499/45766/1/G%c3%bcl%c5%9fah%20%c3%87etindar%c4%b1%20Demirci-.pdf
- See also: Coşkun, A., Arslan, S., & Okcu, G. (2020). Gebe Kadınlarda Gebelik Algısının Stres, Demografik ve Obstetrik Özellikler Açısından İncelenmesi. Journal of Education & Research in Nursing/Hemşirelikte Eğitim ve Araştırma Dergisi, 17(1). — https://jag.journalagent.com/jern/pdfs/JERN-79989-RESEARCH_ARTICLE-COSKUN.pdf
- See also: Boşnak, M., Kurt, A. H., & Yaman, S. (2017). Beynimizin müzik fizyolojisi. Kahramanmaraş Sütçü İmam Üniversitesi Tıp Fakültesi Dergisi, 12(1), 35-44. — https://dergipark.org.tr/tr/download/article-file/322279
- See also: Arkalı, G. T. (2021). Gebelikte Uyku Kalitesi İle Gebelik Uyumu Arasındaki İlişkinin İncelenmesi (Master's thesis, Aydın Adnan Menderes Üniversitesi Sağlık Bilimleri Enstitüsü). — https://tez.yok.gov.tr/UlusalTezMerkezi/tezSorguSonucYeni.jsp
- See also: Akalın A, Şahin S. Preeklampsi: Tanı ve Hemşirelik Yönetiminde Güncel Yaklaşımlar. Journal of Human Rhythm 2018; 4(2): 88-97.) — https://dergipark.org.tr/tr/download/article-file/497288